CLINICAL TRIAL: NCT06655038
Title: A Decent and Healthy Air for Everyone (ADHAirE) : a Randomized Controlled Trial to Improve the Implementation of Tobacco-free School Policies
Brief Title: ADHAirE : a Randomized Controlled Trial to Improve the Implementation of Tobacco-free School Policies
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: FARES (Fonds des affections respiratoires asbl) (Unknown); Observatoire de la santé du Hainaut (Unknown); SEPT (Service d'Etude et de Prévention du Tabagisme) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ADHAIRE
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Smoking; Adolescent Behavior
Keywords: School; Prevention; Advocacy coalition; Social norms
MeSH Terms: conditions — Smoking; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Schools will be the target of an intervention. The 20 participating schools will be randomly assigned either to the intervention arm or to the control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advocacy coalition (Experimental): Feedback + advocacy coalition
  Interventions: Behavioral: Advocacy coalition; Behavioral: Feedback
- Control (Active Comparator): Only feedback
  Interventions: Behavioral: Feedback

INTERVENTIONS:
Behavioral: Advocacy coalition — * set up a task force composed of school stakeholders (students, teachers, educators, principle,...). These stakeholders will meet 4 times a year to improve the implementation and enforcement of TFSP through rules that are accepted, adopted and to which all school actors adhere.
  * share of good practices in implementation with the other schools of the intervention arm through a sharing platform and two annual meetings.
  * support to reffer nicotine-dependant students and staff members to smoking cessation programs.
  * support in the implementation of TFSP and in getting all school actors on board, by the research team, but also by local health promotion partners.
  Arms: Advocacy coalition
Behavioral: Feedback — Feedback on the basis of the audit and the surveys

SUMMARY:
The goal of this cluster randomized controlled trial is to learn if the set up of an advocacy coalition in secondary schools can improve the implementation of tobacco-free school policies (TFSP) to prevent adolescent smoking.

The main questions it aims to answer are:

1. To what extent is an advocacy coalition related to smoking prevention implementable in school's routine ?
2. Is an advocacy coalition an effective way to prevent smoking among adolescents and shift smoking norms in school?

Schools in the intervention arm will be compared to schools in the control arm, to test the effectiness of the advocacy coalition to improve the implementation of TFSP.

Schools in the intervention arm will put in place an advocacy coalition, that is

* Set up a task force composed of school stakeholders (students, teachers, educators, principle,...)
* Share their good practices regarding implementation with the other schools of the intervention arm
* Be supported to reffer nicotine-dependant students and staff members to smoking cessation programs

Continuous evaluation is planned to assess the effectiveness of this intervention.

DETAILED DESCRIPTION:
The ADHAirE project is an experimental study to prevent adolescent smoking.

Its objectives are to

1. Improve the implementation of tobacco-free school policies (TFSP, that is, prohibition of smoking for everyone, anytime, anywhere on the school grounds)
2. Make these TFSP part of school's routine practice
3. Decrease adolescents initiating or reporting smoking

To achieve those goals, schools will put an advocacy coalition in place, that is:

* They wil set up a task force composed of school stakeholders (students, teachers, educators, principle,...). These stakeholders will meet 4 times a year to improve the implementation and enforcement of TFSP through rules that are accepted, adopted and to which all school actors adhere.
* They will share their good practices regarding implementation with the other schools of the intervention arm through a sharing platform and two annual meetings.
* They will be supported to reffer nicotine-dependant students and staff members to smoking cessation programs.
* They will also be supported in the implementation of TFSP and in getting all school actors on board, by the research team, but also by local health promotion partners.

The intervention will be carry out during two years in secondary schools in the Hainaut province, Belgium. This province has one of the highest smoking prevalence in the country and the lowest income level.

A cluster randomized controlled trial will test the effectiveness of the advocacy coalition to improve the implementation of TFSP.

Schools (the clusters) are randomly assigned either to the intervention arm (and set up the advocacy coalition) or to the control arm (and try to achieve the objectives without the advocacy coalition). Randomization will be cross-stratified on the basis of their geographical location (to avoid contamination biases) and social-economic status.

The main questions this study aims to answer are:

1. To what extent is an advocacy coalition related to smoking prevention implementable in school's routine ?
2. Is an advocacy coalition an effective way to prevent smoking among adolescents and shift smoking norms in school?

To answer these questions:

1. We will make an audit on the state of the school policy regarding smoking and tobacco products.
2. A survey will be carried out among staff' members of the participating schools on their engagement in the project, their opinion about smoking prevention at school and their smoking status.
3. A survey will be carried out among adolescents from the 3rd and 4th grade, following a repeated cross-sectional design. Questionnaires will focus on epidemiological indicators such as smoking status and initiation, but also on social norm features such as beliefs and perceptions adolescents hold about smoking.

These evaluations will occur at three times: at baseline, at one year of follow-up and at two years of follow-up. Results of these evaluations will serve to give a feedback to the schools on their situation regarding smoking (regardless to treatment arm to which the school is assigned).

ELIGIBILITY:
These criteria concern adolescents who will take part in the surveys.

Inclusion Criteria:

* student at a secondary school participating in the study
* student of the 3rd and 4th grade

Exclusion Criteria:

* student at a secondary school not participating in the study
* student of another grade than 3rd and 4th grade

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Smoking prevalence | 2 years
  Impact of the advocacy coalition on smoking prevalence and smoking initiation

SECONDARY OUTCOMES:
Smoking norm | 2 years
  Impact of the advocacy coalition on social norms about smoking among adolescents

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Lorant, Professor, Principal Investigator — Université Catholique de Louvain
Locations (1):
- UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laloux P, Melard N, Lorant V. Implementation of school tobacco policies: The advocacy coalition approach. Protocol of the ADHAirE study, a cluster randomized controlled trial. Tob Prev Cessat. 2025 Mar 24;11. doi: 10.18332/tpc/202392. eCollection 2025. PMID 40130233
- See also: Link to the funders' website — https://cancer.be/projets/equipe-du-professeur-vincent-lorant-2022/